CLINICAL TRIAL: NCT04665089
Title: Immunomodulatory Role and Clinical Impact of Erythromycin in Critically Septic Patients: a Randomized Clinical Trial
Brief Title: Erythromycin in Septic Patients: Immunomodulatory Role and Clinical Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Ahlem Trifi, Associate Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rabta
Record Dates: First submitted 2020-11-20; First posted 2020-12-11 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Sepsis; Septic Shock; Immunoinflammatory Response
Keywords: sepsis; erythromycin; immunity; inflammation; mortality
MeSH Terms: conditions — Sepsis; Shock, Septic; Inflammation | interventions — Erythromycin

STUDY DESIGN:
Intervention Model Description: single-blind randomized clinical trial comparing 2 arms: erythromycin versus a placebo
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythromycin arm (Active Comparator): The erythromycin arm (n=55) receives, in addition to the standard antimicrobial therapy, erythromycin 1 g three times per day intravenously: each gram is diluted in 250 ml of 5% glucose serum to be administered over 1 hour for 5 days.
  Interventions: Drug: Erythromycin
- Placebo arm (Placebo Comparator): The placebo arm (n=55) receives, in addition to the standard antimicrobial therapy, isotonic saline, intravenously, 20 ml diluted in 250 ml of 5% glucose serum to be administered over 1 hour for 5 days.
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin — Before each intervention (either at inclusion: day 0) and after the end of 5 days of erythromycin or placebo (day 6), the following dosages will be performed:
  * Pro-inflammatory cytokine (TNF alpha)
  * Anti-inflammatory cytokine (IL-10)
  * Procalcitonin (PCT) Then, analysis of the variations in the TNF/ IL-10 ratio, the blood count, CRP and PCT parameters (between Day 0 and Day 6)
  Other Names: specific dosages

SUMMARY:
In sepsis and septic shock, the host response is characterized by a complex of immune-inflammatory reactions; triggered and activated by microbial components. These reactions are controlled by a balance of pro-inflammatory cytokines and anti-inflammatory cytokines. The imbalance of this immune response is a source of organ dysfunction; major prognostic factor during septic condition. This pretext has created the need for therapies aimed to modulate the overstated of host response. During the past 2 decades, macrolide molecules proved interest to be immunomodulatory agents; due beyond their antibacterial activity. Their regulatory role in the production of cytokines was demonstrated in the management of severe acute community pneumonia.

The investigators hypothesize that the adjunction of macrolides to standard therapy in patients with sepsis or septic shock is associated to a favorable immunomodulatory and clinical effects.

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. It is considered as the main cause of death in critically ill patients ranging from 20 to 50%. These alarming death rates have prompted several intense research efforts to better understand the mechanisms underlying the pathogenesis of sepsis. Currently, sepsis is recognized as a complex entity created by an immuno-inflammatory reaction of the infected host; triggered and activated by microbial components. This reaction brings together the cellular and humoral immunity defense systems. Activation of the cellular system involves macrophages, polymorphonuclear cells, lymphocytes and endothelial cells.

Therefore, pro-inflammatory cytokines are secreted in order to control the infection (IL-1, IL-6, IL-8, and TNF-alpha). Simultaneously, anti-inflammatory cytokines (IL-4, IL-10) are also released, allowing a local and systemic regulation of the inflammatory cascade. The imbalance of this immune response is a source of organ dysfunction aggravated by the lack of tissue oxygenation.

Understanding that sepsis results from a disproportionate immune-inflammatory response have created the need for therapies aimed to modulate the overstated host response. The agents tested were: anti-endotoxin antibodies, tumor necrosis factor (TNF), anti-TNF-alpha, recombinant human activated protein C (rhAPC), stress-dose hydrocortisone and statins. Most of these clinical trials showed no obvious clinical impact or a limited clinical efficacy.

During the past 2 decades, macrolides molecules were revealed to be immune-modulator agents; beyond their antibacterial activity. Their immune-modulator properties result from their ability to induce the activity of various immune cells and their regulatory role in the production of cytokines. Several cellular targets and mechanisms have been described to explain the immune-modulator effects of macrolides: Respiratory epithelial cells and innate immunity cells. Overall, macrolides decrease the production of pro-inflammatory cytokines by innate and adaptive immunity cells.

In this clinical trial, the investigators are focusing on the effects of macrolides on the pro-inflammatory / anti-inflammatory balance by assaying cytokines and other immune-inflammatory markers during sepsis and septic shock. The main hypothesis is that the use of macrolides in addition to standard therapy in critically septic patients has a favorable immune-modulator and clinical effects compared to critically septic patients not receiving macrolide.

ELIGIBILITY:
Inclusion Criteria:

* a patient in whom the diagnosis of sepsis or septic shock is diagnosed (According to the definitions updated by the sepsis 3 consensus in 2016)

Exclusion Criteria:

* Macrolide use for another indication.
* Known allergy to macrolides.
* A corrected QT prolonged (> 440 ms for man and 460 ms for woman) or taking drugs with an increased risk of QT prolongation.
* QT prolongation attributed to erythromycin
* Underlying dysimmunity (unbalanced diabetes, autoimmune disease, etc.)
* Pregnant or breastfeeding woman.
* Death or discharge while participating in the protocol (day 0 to day 6)
* Non-compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change of TNF α / IL-10 ratio | Change from Baseline TNF α / IL-10 ratio at 6 days
  The pro-inflammatory / anti-inflammatory balance will be estimated by measuring the TNF α / IL-10 ratio at baseline and that at day 6. The difference (Δ) of TNF α / IL-10 ratio between day 0 (or baseline) and day 6 will be calculated in each arm then compared between the 2 arms.

SECONDARY OUTCOMES:
mortality | 28 days
  28-day mortality
Procalcitonine | At day 0 and day 6 of inclusion
  bilogical parameter with measurement of the difference (Δ) in procalcitonine between day 6 and day 0
vasopressors requirement in mg/H | during follow-up, an average of 28 days
  maximum dose of vasopressors use
vasopressors requirement in days | during follow-up, an average of 28 days
  time needed of vasopressors use

CONTACTS AND LOCATIONS:
Locations (1):
- intensive care unit of the University Hospital Center La Rabta, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trifi A, Tlili B, Kallel Sellami M, Feki M, Mehdi A, Seghir E, Messaoud L, Abdellatif S, Ben Lakhal S. Immunologic effect and clinical impact of erythromycin in septic patients: A randomized clinical trial. J Crit Care. 2024 Jun;81:154533. doi: 10.1016/j.jcrc.2024.154533. Epub 2024 Feb 14. PMID 38359518